CLINICAL TRIAL: NCT06054685
Title: A Study on the Association Between Body Composition and Survival in Digestive System Tumors and Immune Treatment Response
Brief Title: Association Between Body Composition and Digestive System Cancer Survival
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-SR-339
Record Dates: First submitted 2023-09-19; First posted 2023-09-26 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Digestive System Cancer
MeSH Terms: conditions — Digestive System Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Routine Clinical Blood Tests
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Investigators intend to utilize clinical data from the Department of Oncology at Jiangsu Provincial People's Hospital to analyze changes in body composition in digestive system tumor patients before and after receiving anti-tumor drug treatment. Investigators aim to uncover the association between baseline body composition and overall/progression-free survival in patients with digestive system tumors. Additionally, Investigators plan to investigate the relationship between changes in body composition during anti-tumor drug treatment (chemotherapy and immunotherapy) and the prognosis of tumor patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged between 18 and 85 years old.
* Patients with histologically confirmed digestive tract cancers, such as esophageal cancer, gastric cancer, small intestinal cancer, colorectal cancer, as well as pancreatic cancer, liver cancer, gallbladder cancer, etc.
* Patients admitted for anti-tumor-related drug treatment.
* Expected survival period of more than three months.
* ECOG PS score: < 4.
* No severe psychological disorders, physical disabilities, dementia, Alzheimer's disease, pulmonary tuberculosis, HIV/AIDS, or other infectious diseases.
* Patients must have sufficient organ and bone marrow function, meeting the following criteria:

  1. Hematological criteria:

     Hemoglobin (Hb) ≥ 90 g/L (without blood transfusion in the past 28 days). Absolute neutrophil count (ANC) ≥ 1.5×109/L. Peripheral blood monocytes > 1500mm3. Platelet count (PLT) ≥ 100×109/L.
  2. Biochemical criteria:

     Total bilirubin (TBIL) ≤ 1.5 × the upper limit of normal (ULN). ALT and AST ≤ 2.5×ULN; if there is liver metastasis, ALT and AST ≤ 5×ULN. Creatinine (Cr) ≤ 1.5×ULN or creatinine clearance rate (CCr) ≥ 60 ml/min (Cockcroft-Gault formula).
  3. Coagulation function is sufficient, defined as international normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 × ULN.
* Women of childbearing potential must have a negative pregnancy test (serum or urine) within seven days before enrollment and must voluntarily use appropriate contraception methods during the observation period and within six months after the last dose.
* Signed informed consent.

Exclusion Criteria:

* Female patients who are pregnant or breastfeeding.
* Patients with accompanying diseases, as judged by the investigator, pose a serious risk to patient safety or may affect the patient's ability to complete the study.
* Patients with poor compliance who refuse to undergo body composition measurements.
* Patients who experience a severe adverse event judged by the investigator as no longer suitable for continued participation in the study or those who become unexpectedly pregnant.
* Patients who are unwilling to continue in the clinical trial and insist on withdrawal.
* The investigator deems it necessary to terminate the study.
* Patients who were mistakenly included but did not meet the criteria.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This prospective study includes digestive system tumor patients treated in the elderly comprehensive ward of Jiangsu Provincial People's Hospital from April 2023 to September 2024. Baseline surveys were conducted between April and May 2023 and between September and October 2024.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-04-17 (Actual); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
PFS | 2025-01-30
  Progress free survival

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No